CLINICAL TRIAL: NCT01416194
Title: COHORT STUDY OF VENOUS THROMBOEMBOLISM AND OTHER CLINICAL ENDPOINTS AMONG OSTEOPOROTIC WOMEN PRESCRIBED BAZEDOXIFENE, BISPHOSPHONATES OR RALOXIFENE IN EUROPE
Brief Title: Bazedoxifene Post Approval Safety Study (PASS) in the European Union (EU)
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1781044
Record Dates: First submitted 2011-08-11; First posted 2011-08-12 (Estimated); Results first posted 2020-05-18 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — bazedoxifene; Diphosphonates; Raloxifene Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Bazedoxifene
  Interventions: Drug: Bazedoxifene
- Primary Comparator
  Interventions: Drug: Bisphosphonate
- Secondary Comparator
  Interventions: Drug: Raloxifene

INTERVENTIONS:
Drug: Bazedoxifene — Patients receiving Bazedoxifene in usual clinical care. In this non-interventional study there is no protocol mandated drug assignment or dosing schedule.
  Groups: Bazedoxifene
Drug: Bisphosphonate — Patients receiving Bisphosphonates in usual clinical care. In this non-interventional study there is no protocol mandated drug assignment or dosing schedule.
  Groups: Primary Comparator
Drug: Raloxifene — Patients receiving Raloxifene in usual clinical care. In this non-interventional study there is no protocol mandated drug assignment or dosing schedule.
  Groups: Secondary Comparator

SUMMARY:
This observational cohort study is being conducted to further characterize selected adverse events of interest among a patient population with osteoporosis who are prescribed bazedoxifene, raloxifene, or a bisphosphonate in usual clinical care outside of a randomized clinical trial setting. The study will compare the rates of the selected clinical events among the three treatment groups.

DETAILED DESCRIPTION:
All women in the database meeting the inclusion criteria will be included in the study without any statistical sampling.

ELIGIBILITY:
Inclusion Criteria:

* Female
* At least one prescription for bazedoxifene, raloxifene, or any bisphosphonate during the study inclusion period (index prescription);
* A recoded diagnosis code of osteoporosis on or within 60 days prior to the index prescription date;
* Age >=45 at the date of the index prescription; and
* At least 6-months of follow-up data in the electronic medical record system prior to the date of the index prescription

Exclusion Criteria:

* There is no exclusion criteria. All women in the database who meet the inclusion criteria will be studied.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women aged 45 or over who have records of receiving bazedoxifene, bisphosphonates or raloxifene in the Cegedim database in Italy and Spain.
Sampling Method: Non-Probability Sample
Enrollment: 10497 (Actual)
Dates: Start 2011-07-25 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1781044&StudyName=Bazedoxifene%20Post%20Approval%20Safety%20Study%20%28PASS%29%20in%20the%20European%20Union%20%28EU%29

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a retrospective, observational, non-interventional study. Data was collected from proprietary longitudinal patient databases (LPD).
Pre-assignment Details: The index date for each participant was the date of first recorded prescription for bazedoxifene, raloxifene or bisphosphonate. Follow-up period was from index date to first incident of primary event or date of last contact, whichever occurred first. Follow-up was maximum up to approximately of 92.1 months.
Groups:
- Bazedoxifene: Participants with postmenopausal osteoporosis received bazedoxifene in usual routine clinical care per summary of product characteristics (SmPC) and dose was adjusted by physicians solely according to medical and therapeutic necessity.
- Raloxifene: Participants with postmenopausal osteoporosis received raloxifene in usual routine clinical care per SmPC and dose was adjusted by physicians solely according to medical and therapeutic necessity.
- Bisphosphonate: Participants with postmenopausal osteoporosis received bisphosphonate in usual routine clinical care per SmPC and dose was adjusted by physicians solely according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Started | 1111 | 2720 | 6666
Completed | 1111 | 2720 | 6666
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set included all women participants in database who met the inclusion criteria and whose data was observed in the study.
Groups:
- Bazedoxifene: Participants with postmenopausal osteoporosis received bazedoxifene in usual routine clinical care per SmPC and dose was adjusted by physicians solely according to medical and therapeutic necessity.
- Total: Total of all reporting groups
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate | Total
Number analyzed (Participants) | 1111 | 2720 | 6666 | 10497
Age, Customized [Count of Participants; unit: Participants]
  From 45-49 years | 51 | 78 | 88 | 217
  From 50-59 years | 479 | 665 | 915 | 2059
  From 60-69 years | 382 | 1229 | 1915 | 3526
  From greater than equal to (>=) 70 years | 199 | 748 | 3748 | 4695
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1111 | 2720 | 6666 | 10497
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Cumulative Incidence of Venous Thromboembolism (VTE)
Description: VTE is defined as deep vein thrombosis (DVT), pulmonary embolism (PE), retinal vein thrombosis, and sinus thrombosis. DVT: occurs when a blood clot forms in a vein located deep inside the body. PE: a blockage of an artery in the lungs by a substance that has moved from elsewhere in the body through the bloodstream (embolism). Sinus thrombosis: presence of a blood clot in the dural venous sinuses, which drain blood from the brain. Retinal vein thrombosis: blockage of the small veins that carry blood away from the retina. Cumulative incidence was calculated as total participants with VTE events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 1.5 [1.0 to 2.4] | 2.2 [1.7 to 2.8] | 4.6 [4.1 to 5.1]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; The hazard ratio from Cox proportional hazard regression models was used for comparison of event rates of the primary and secondary endpoints in each treatment group. Statistical two-sided tests was used with a significance level of 0.05; Test type: Superiority; p < 0.01, Regression, Logistic; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.3 to 0.7]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.91, Regression, Logistic; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.4 to 2.2]

2. Secondary Outcome: Cumulative Incidence of Ischemic Stroke
Description: Ischemic stroke is caused by a blockage in an artery that supplies blood to the brain. Cumulative incidence was calculated as total participants with ischemic stroke events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 2.2 [1.5 to 3.2] | 2.6 [2.1 to 3.3] | 6.7 [6.2 to 7.4]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, Regression, Logistic; Hazard Ratio (HR) = 0.5, 95% CI 2-sided [0.3 to 0.7]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.76, Regression, Logistic; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.5 to 2.4]

3. Secondary Outcome: Cumulative Incidence of Cardiac Disorders
Description: Cardiac disorders included myocardial infarction, myocardial ischemia, and coronary occlusion. Cumulative incidence was calculated as total participants with cardiac disorders events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 2 [1.3 to 3.0] | 3 [2.4 to 3.7] | 6.6 [6.1 to 7.3]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.01, Regression, Logistic; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.3 to 0.9]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.37, Regression, Logistic; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.4 to 1.5]

4. Secondary Outcome: Cumulative Incidence of Atrial Fibrillation
Description: Atrial fibrillation is an irregular heartbeat that increases the risk of stroke and heart disease. Cumulative incidence was calculated as total participants with atrial fibrillation events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 2.8 [2.0 to 3.9] | 4.3 [3.6 to 5.1] | 6.5 [6.0 to 7.2]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.10, Regression, Logistic; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.5 to 1.1]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.19, Regression, Logistic; Hazard Ratio (HR) = 0.7, 95% CI 2-sided [0.4 to 1.2]

5. Secondary Outcome: Cumulative Incidence of Biliary Events
Description: Biliary events included cholecystitis and cholelithiasis. Cumulative incidence was calculated as total participants with biliary events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 1.8 [1.2 to 2.8] | 2 [1.6 to 2.6] | 4 [3.5 to 4.5]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, Regression, Logistic; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.3 to 0.7]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.90, Regression, Linear; Hazard Ratio (HR) = 1.0, 95% CI 2-sided [0.4 to 2.1]

6. Secondary Outcome: Cumulative Incidence of Hypertriglyceridemia
Description: Hypertriglyceridemia refers to high blood levels of triglycerides. Cumulative incidence was calculated as total participants with hypertriglyceridemia events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 9.7 [8.1 to 11.6] | 10.6 [9.5 to 11.8] | 6 [5.4 to 6.5]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, Regression, Logistic; Hazard Ratio (HR) = 1.9, 95% CI 2-sided [1.4 to 2.5]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.74, Regression, Logistic; Hazard Ratio (HR) = 0.9, 95% CI 2-sided [0.7 to 1.3]

7. Secondary Outcome: Cumulative Incidence of Clinical Fractures
Description: A fracture is a break in a bone. Cumulative incidence was calculated as total participants with clinical fractures events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 4.4 [3.4 to 5.8] | 8.2 [7.3 to 9.3] | 12.8 [12.0 to 13.6]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, Regression, Logistic; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.3 to 0.6]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.01, Regression, Logistic; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.4 to 0.9]

8. Secondary Outcome: Cumulative Incidence of Renal Failure
Description: Cumulative incidence was calculated as total participants with renal failure events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 0.8 [0.4 to 1.5] | 2.3 [1.8 to 3.0] | 4.8 [4.3 to 5.3]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, Regression, Linear; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.1 to 0.5]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.06, Regression, Linear; Hazard Ratio (HR) = 0.4, 95% CI 2-sided [0.2 to 1.1]

9. Secondary Outcome: Cumulative Incidence of All Malignancies
Description: All malignancies included and not limited only to thyroid, breast, renal, genital / urogenital, lung cancer, gastrointestinal tract and respiratory tract. Cumulative incidence was calculated as total participants with malignancies events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 3.2 [2.3 to 4.3] | 4.4 [3.7 to 5.2] | 6.6 [6 to 7.2]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, Regression, Linear; Hazard Ratio (HR) = 0.5, 95% CI 2-sided [0.3 to 0.7]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.38, Regression, Linear; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.5 to 1.4]

10. Secondary Outcome: Cumulative Incidence of Different Types of Malignancies
Description: In this outcome measure, cumulative incidence of different types of malignancies included breast, renal, thyroid, genital / urogenital, gastrointestinal tract, lung and respiratory tract were calculated. Cumulative incidence for each type of malignancy was calculated as total participant with the respective malignancy events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence for each type of malignancy was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants
  Malignancies - Thyroid: number analyzed (Participants) | 0 | 2720 | 6666
  Malignancies - Thyroid |  | 0.1 [0 to 0.3] | 0.2 [0.1 to 0.3]
  Malignancies - Breast | 0.4 [0.1 to 0.9] | 0.6 [0.4 to 1.0] | 1.4 [1.1 to 1.7]
  Malignancies - Renal: number analyzed (Participants) | 0 | 2720 | 6666
  Malignancies - Renal |  | 0.1 [0.0 to 0.3] | 0.1 [0.0 to 0.2]
  Malignancies - Genital / Urogenital | 0.5 [0.2 to 1.2] | 0.4 [0.2 to 0.7] | 0.5 [0.3 to 0.7]
  Malignancies - Lung | 0.3 [0.1 to 0.8] | 0.4 [0.2 to 0.7] | 0.3 [0.2 to 0.5]
  Malignancies- Gastrointestinal | 1.1 [0.6 to 1.9] | 1.1 [0.8 to 1.6] | 1.5 [1.2 to 1.8]
  Malignancies- Respiratory: number analyzed (Participants) | 1111 | 0 | 6666
  Malignancies- Respiratory | 0.1 [0.0 to 0.5] |  | 0.1 [0.0 to 0.2]

11. Secondary Outcome: Cumulative Incidence of Depression
Description: Cumulative incidence was calculated as total participants with depression events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 10.1 [8.4 to 12.0] | 9.2 [8.2 to 10.4] | 8.6 [7.9 to 9.3]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.24, Regression, Linear; Hazard Ratio (HR) = 1.2, 95% CI 2-sided [0.9 to 1.5]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.59, Regression, Linear; Hazard Ratio (HR) = 1.1, 95% CI 2-sided [0.8 to 1.6]

12. Secondary Outcome: Cumulative Incidence of Selected Ocular Events
Description: Selected ocular events included retinal vascular occlusions, disorders of the globe, iris, ciliary body, retina, eye adnexa and cornea. Cumulative incidence was calculated as total participants with selected ocular events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 8 [6.6 to 9.8] | 12.5 [11.3 to 13.8] | 10.8 [10.1 to 11.6]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.03, Regression, Logistic; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.6 to 1.0]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.19, Regression, Linear; Hazard Ratio (HR) = 0.8, 95% CI 2-sided [0.6 to 1.1]

13. Secondary Outcome: Cumulative Incidence of Thyroid Disorders- Goitre
Description: Goitre is a swelling in the neck resulting from an enlarged thyroid gland. Cumulative incidence was calculated as total participants with thyroid disorders-goitre events during follow-up period divided by total persons at risk during follow-up period*100 and hence cumulative incidence was expressed as percentage of participants.
Time Frame: Up to a maximum of follow-up period of 92.1 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bazedoxifene | Bisphosphonate | Raloxifene
Number analyzed (Participants) | 1111 | 2720 | 6666
percentage of participants | 1.6 [1.0 to 2.5] | 2.5 [1.9 to 3.1] | 3.8 [3.4 to 4.3]
Statistical Analysis 1: Comparison: Bazedoxifene vs Bisphosphonate; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.01, Regression, Linear; Hazard Ratio (HR) = 0.3, 95% CI 2-sided [0.2 to 0.5]
Statistical Analysis 2: Comparison: Bazedoxifene vs Raloxifene; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.24, Regression, Linear; Hazard Ratio (HR) = 0.6, 95% CI 2-sided [0.3 to 1.3]

ADVERSE EVENTS:
Time Frame: Not applicable as safety data was not planned to be collected during the study
Description: Safety data was not planned to be collected during the study.
Arm/Group | Bazedoxifene | Raloxifene | Bisphosphonate
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2013-08-19): https://cdn.clinicaltrials.gov/large-docs/94/NCT01416194/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-27): https://cdn.clinicaltrials.gov/large-docs/94/NCT01416194/SAP_001.pdf